CLINICAL TRIAL: NCT00982527
Title: Intraoperative Fenoldopam Infusion in Children Requiring Cardiopulmonary Bypass During Cardiac Surgery
Brief Title: Fenoldopam in Pediatric Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Zaccaria Ricci, medical doctor, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSCPB-1
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Kidney Failure, Acute
Keywords: cardiopulmonary bypass; pediatric cardiac surgery; acute renal failure; renal biomarkers; fenoldopam; Focus on optimization of perfusion during pediatric CPB
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Chloride; Fenoldopam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline blinded infusion
  Interventions: Drug: Placebo; Drug: Fenoldopam
- Fenoldopam (Active Comparator): Drug infusion
  Interventions: Drug: Placebo; Drug: Fenoldopam

INTERVENTIONS:
Drug: Placebo — Saline continuous infusion during cardiopulmonary by pass at 1 ml/h
  Other Names: saline
Drug: Fenoldopam — Fenoldopam continuous infusion at 1 mcg/kg/min during cardiopulmonary bypass. Infusion preparation is mad in order to match the rate 1 ml/h of placebo infusion.
  Other Names: corlopam

SUMMARY:
The purpose of this study is to determine whether fenoldopam infusion during cardiopulmonary bypass in young children with congenital heart disease is able to reduce indicators of acute kidney injury (biomarkers reduction, diuresis increase) compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital heart disease, less than one year old, undergoing surgery with the use of cardiopulmonary bypass

Exclusion Criteria:

* Children over one year old, correction for ventricular or atrial septal defect, need for deep hypothermic circulatory arrest, preoperative renal dysfunction.

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Reduction of urinary and/or serum levels of biomarker NGAL in treated group versus controls | End of surgery and 12 hours postoperatively

SECONDARY OUTCOMES:
Reduction of urinary and/or serum levels of cystatin C, increase of diuresis and improvement of perfusion markers in treated group versus controls | End of surgery and 12 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Zaccaria Ricci, MD, Principal Investigator — Bambino Gesu Hospital; Sergio Picardo, MD, Study Director — Bambino Gesù Hospital
Locations (1):
- Bambino Gesù Hospital, Rome, Lazio, Italy

REFERENCES:
- [Background] Dent CL, Ma Q, Dastrala S, Bennett M, Mitsnefes MM, Barasch J, Devarajan P. Plasma neutrophil gelatinase-associated lipocalin predicts acute kidney injury, morbidity and mortality after pediatric cardiac surgery: a prospective uncontrolled cohort study. Crit Care. 2007;11(6):R127. doi: 10.1186/cc6192. PMID 18070344
- [Background] Ricci Z, Stazi GV, Di Chiara L, Morelli S, Vitale V, Giorni C, Ronco C, Picardo S. Fenoldopam in newborn patients undergoing cardiopulmonary bypass: controlled clinical trial. Interact Cardiovasc Thorac Surg. 2008 Dec;7(6):1049-53. doi: 10.1510/icvts.2008.185025. Epub 2008 Sep 9. PMID 18782787
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014
- [Derived] Ricci Z, Luciano R, Favia I, Garisto C, Muraca M, Morelli S, Di Chiara L, Cogo P, Picardo S. High-dose fenoldopam reduces postoperative neutrophil gelatinase-associated lipocaline and cystatin C levels in pediatric cardiac surgery. Crit Care. 2011 Jun 29;15(3):R160. doi: 10.1186/cc10295. PMID 21714857